CLINICAL TRIAL: NCT03441139
Title: Randomized Controlled Multicenter Prospective Open-label Study of the Efficacy of the Percutaneous Cryotherapy Combined or Not With a Medical Analgesia in the Treatment of Patients With Uncontrolled Painful Musculoskeletal Metastasis
Brief Title: Efficacy of Cryotherapy Combined or Not With Analgesics in Uncontrolled Painful Musculoskeletal Metastasis
Acronym: CRYO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty to recruit patient.
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ET17-016 (Cryoanalgesia)
Record Dates: First submitted 2018-01-29; First posted 2018-02-22 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Musculoskeletal Pain
Keywords: Randomized controlled trial; Musculoskeletal metastasis; Cancer pain; Percutaneous cryotherapy; Medical supportive care
MeSH Terms: conditions — Musculoskeletal Pain; Cancer Pain | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy + medical analgesics (Experimental): Percutaneous Cryotherapy and medical analgesics according to the investigator's discretion
  Interventions: Other: Cryotherapy + Medical analgesics
- Medical analgesics (Active Comparator): Medical analgesics alone according to the investigator's discretion
  Interventions: Drug: Medical Analgesics

INTERVENTIONS:
Other: Cryotherapy + Medical analgesics — Percutaneous cryotherapy: A complete cycle of treatment will require 2 freezing 10-minutes periods, separate by a 9-minutes passive and 1-minute active thaw, with the cryoablation system. Dimension of the iceball coverage above the tumor will be monitored by non-contrast CT or MRI during the freezing cycle.
  Medical supportive care: Best analgesic therapy at investigator's discretion
  Other Names: Percutaneous cryotherapy + Medical analgesics
  Arms: Cryotherapy + medical analgesics
Drug: Medical Analgesics — Best analgesic therapy at investigator's discretion
  Other Names: Best medical medical analgesics
  Arms: Medical analgesics

SUMMARY:
The primary objective of this trial is to compare the efficacy of 2 analgesic strategies, based on percutaneous cryotherapy plus medical supportive care versus medical supportive care alone in the treatment of cancer patients with painful musculoskeletal metastasis.

DETAILED DESCRIPTION:
There is a substantial body of evidences that support the rationale for percutaneous cryotherapy in the treatment of painful musculoskeletal metastasis. Since the available results are based exclusively on retrospective and single-arm prospective studies, all authors agree that preliminary data deserves further investigation to provide high level evidences.

Current knowledge, along with the need for relieving patients' pain, already leads interventional radiologists to introduce analgesic cryotherapy in their routine practice. Our team usually notes a clinically significant pain relief that is immediate, continuous and prolonged in these patients. However, facing the lack of comparative studies, this technique is still proposed to patients with poor life-expectancy.

Percutaneous cryotherapy is an innovative strategy in the treatment of patients with uncontrolled painful metastases. It could provide a significant and durable pain relief and a better quality of life, earlier in the patient's care pathway.

The study group hypotheses that an early procedure of percutaneous cryotherapy is able to provide painful patients with better and prolonged analgesia and quality of life.

A prospective controlled study is proposed with two analgesic strategies (percutaneous cryotherapy plus medical supportive care versus medical supportive care alone) in patients with a painful metastasis not controlled by conventional analgesia strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the day of consenting to the study;
* Patient with at least 1 painful metastasis with a musculoskeletal involvement;
* Patient referred to a Pain Management Unit to optimize the analgesic strategy;
* Painful metastatic lesion that fulfils with all the following :

  * Pain must be correlated with an identifiable lesion on imaging (Computed Tomography, Magnetic Resonance Imaging or Ultrasonography)
  * Level of mean pain within the past 24 hours of at least 4/10 (numeric rating scale)
  * Painful metastasis suitable for a procedure of percutaneous cryotherapy
* Life-expectancy longer than 6 months;
* Performance Status of the ECOG ≤2;
* Neutrophils count > 1 Gi/l within the past 14 days;
* Adequate coagulation panel (as per the investigator judgement);
* Ability to understand and willingness for follow-up visits;
* Covered by a medical insurance;
* Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrolment.

Exclusion Criteria:

* Patient with a primary tumor of leukemia, lymphoma or myeloma;
* Tumor involving a weight bearing long bone of the lower limbs with the tumor causing more than 50% of cortical bone;
* Lesion amenable to any curative intervention;
* Formal indication for local analgesic procedure other than percutaneous cryotherapy;
* Prior radiotherapy on the targeted lesion within the 3 weeks prior to randomization;
* Patient with any contraindication for the procedure of percutaneous cryotherapy, including treatment requiring ice ball formation within 0.5 cm of the spinal cord, brain, other critical nerve, structure, large abdominal vessels such as the aorta or inferior vena cava, bowel or bladder (except if active or passive thermic protection can be performed);
* Uncontrolled coagulopathy or bleeding disorders;
* Evidence of pregnancy, breast-feeding, or patient wishing to become pregnant during the study;
* Active, uncontrolled infection;
* Any cognitive impairment or any disease that may restrain the use of numeric scales and the administration of quality of life questionnaires;
* Clinically significant unrelated systemic illness (e.g., serious infection or significant cardiac, pulmonary, hepatic, or other organ dysfunction) that would likely interfere with study procedures or results;
* Concurrent participation in other experimental studies that could interfere with the primary endpoint assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Time to analgesic strategy failure | Time from the date of randomization to the date of analgesic strategy failure assessed up to 6 months
  Failure will be defined as at least, one of the following situations: Reescalation of the mean local pain by 2 points or more from the lowest pain score from baseline; Absence of pain relief ≥ 2 points 3 months after randomization; Indication of any other loco regional analgesic procedure (radiotherapy, interventional radiology or surgery).

SECONDARY OUTCOMES:
Percentage of pain relief | Weekly for the first 3 months, then monthly assessed up to 6 months
  Percentage of pain relief from baseline, rated by patients
Depth of local pain relief | Numeric rating scale (scale range from 0 [no pain] to 10 [worst imaginable pain]): Weekly for the first 3 months, then monthly assessed up to 6 months
  Evaluation using the numeric rating scale
Depth of local pain relief | Brief Pail Inventory : Monthly assessment up to 6 months
  Evaluation using the Brief Pain Inventory
The impact of local pain on the patient's quality of life | Monthly assessment up to 6 months
  Using the FACT-BP questionnaire
The impact of local pain on the patient's quality of life | Monthly assessment up to 6 months
  Using the EuroQOL-5Dimensions-5Levels questionnaire
Description of analgesic consumption | Weekly for the first 3 months, then monthly assessed up to 6 months
  Using a booklet completed by the patients and/or the investigator
Overall Survival | From date of randomization to date of death from any cause or date of LPLV (estimated date: March 2020)
  Time from the date of randomization to the date of death due to any cause
Tolerance profile | Date of last visit (Month 6 +/- 28 days)
  Tolerance assessed according to the NCI-CTC AE version 4

OTHER OUTCOMES:
Cost-effectiveness analysis | Date of last visit (Month 6 +/- 28 days)
  All the resources consumption will be collected during the 6-months timeframe: Hospitalization costs (outpatient, inpatient, and home care), external consultations and wider examinations (eg MRI), transportation costs.
Cost-utility analysis | Date of last visit (Month 6 +/- 28 days)
  All the resources consumption will be collected during the 6-months timeframe: Hospitalization costs (outpatient, inpatient, and home care), external consultations and wider examinations (eg MRI), transportation costs.
Budget impact analyses | One-year baseline period. Will be performed in case the experimental strategy dominates the standard strategy
  Quantication of financial consequences of rolling out the innovative strategy throughout the health system (i.e. the replacement of Medical supportive care by Medical supportive care + Percutaneous cryotherapy)

CONTACTS AND LOCATIONS:
Overall Officials: Charles MASTIER, MD, Principal Investigator — Centre Leon Berard
Locations (8):
- France (8):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancérologie de Montpellier-Val d'Aurelle, Montpellier
  - Institut de Cancérologie de l'Ouest - Centre René Gauducheau, Saint-Herblain
  - Institut Paul Strauss, Strasbourg
  - CHRU de Strasbourg, Strasbourg
  - Institut Gustave Roussy, Villejuif